CLINICAL TRIAL: NCT03375086
Title: A Phase 1 Study of APX3330 in Patients With Advanced Solid Tumors
Brief Title: A Study of APX3330 in Patients With Advanced Solid Tumors
Acronym: APX3330
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apexian Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX_CLN_0011
Record Dates: First submitted 2017-11-21; First posted 2017-12-15 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — E 3330

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center, dose escalation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Patients will receive APX3330 orally, twice per day until disease progression
  Interventions: Drug: APX3330

INTERVENTIONS:
Drug: APX3330 — APX3330 will be supplied as 60 and 120 mg orally administered tablets. Patients will receive a fixed dose of APX3330 twice daily (i.e., bid) each day of a 21-day cycle. The starting dose of APX3330 will be a daily dose of 240 mg (i.e., 120 mg/dose bid). Doses will be increased until identification of a maximum tolerated dose or bio-effective dose, whichever is lower.
  Other Names: E3330

SUMMARY:
This is a Phase 1, multi-center, open-label, dose-escalation oncology study of APX3330 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Apurinic/apyrimidinic endonuclease 1/redox factor-1 (APE1/Ref-1) is a protein that regulates multiple transcription factors involved in cancer cell signaling and APX3330 is a highly selective inhibitor of APE1/Ref-1 redox function.

The anti-tumor effect of APX330 has been demonstrated in a variety of preclinical models and the human safety profile of APX3330 was established in prior clinical studies. Apexian Pharmaceuticals is developing APX3330 as an orally administered anti-cancer agent targeting the APE1/Ref-1 protein.

APX_CLN_0011 is a Phase 1, multi-center, open-label, dose-escalation oncology study in patients with advanced solid tumors. The study primary objective is to determine the recommended Phase 2 study dose of APX3330. Secondary objectives include assessment of APX3330 safety, anti-tumor activity, pharmacokinetic and pharmacodynamic profile.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from the patient.
2. Patient must be > 18 years of age.
3. Patient must have recurrent or advanced cancer (i.e., solid tumors) for whom standard therapy offers no curative potential.
4. Evaluable disease by RECIST v1.1.
5. Performance status (PS) of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale. Note: PS 2 patients can only participate if, in the assessment of the clinical investigator, and with the consent of the medical monitor, the patient has the ability to participate in the clinical study for a minimum of at least 2 cycles.
6. > 21 days from therapeutic radiation or chemotherapy (>6 weeks from nitrosoureas and mitomycin C) and recovery to (NCI CTCAE v4.03) Grade ≤ 1 from all clinically significant toxicities related to prior therapies.
7. Must have adequate organ function defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
   2. Platelet ≥ 100 x 10^9/L.
   3. Hemoglobin ≥ 9 g/dL.
   4. Activated partial thromboplastin time/ partial thromboplastin time (aPTT/PTT) ≤ 1.5 x ULN
   5. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN). In the case of known (i.e., radiological or biopsy documented) liver metastasis, serum transaminase levels must be < 5 x ULN.
   6. Total serum bilirubin ≤ 1.5 x ULN, (except for patients with known Gilbert's Syndrome ≤ 3 x ULN is permitted)
   7. Renal: Serum creatinine < 2.0 x ULN or creatinine clearance ≥ 50 mL/min/1.73m^2 for patients with serum creatinine levels above 2 x ULN.
8. Agreement to use acceptable methods of contraception during the study and for at least 120 days after the last dose of APX3330 if sexually active and able to bear or beget children.

Exclusion Criteria:

1. Diagnosed with another malignancy within the past 2 years (excluding a history of carcinoma in situ of the cervix, superficial non-melanoma skin cancer, superficial bladder cancer, or endometrial cancer that has been adequately treated, or stage 1 prostate cancer that does not require treatment).
2. History of a major surgical procedure or a significant traumatic injury within 14 days prior to commencing treatment, or the anticipation of the need for a major surgical procedure during the course of the study.
3. Patients who have been treated with an investigational agent within 21 days prior to the first dose of study drug.
4. Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, New York Heart Association (NYHA) class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, active hepatitis B, C or HIV, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.
5. Impaired liver function Child-Pugh class B or C (score 7-15).
6. Women who are pregnant or lactating.
7. Patients with evidence of symptomatic brain metastases. Patients with treated (surgically excised or irradiated) and stable brain metastases are eligible assuming the patient has adequately recovered from treatment, the treatment was at least 28 days prior to initiation of study drug, and baseline brain computed tomography (CT) with contrast, or magnetic resonance imaging (MRI) within 14 days of initiation of study drug, is negative for new or worsening brain metastases
8. Other concurrent chemotherapy, immunotherapy, radiotherapy or investigational therapy except for hormonal therapy (e.g., tamoxifen, etc.).
9. Patients requiring palliative radiotherapy to lesions that are defined as target lesions by RECIST criteria at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 12 months
  Identification of the safety and tolerability of APX3330

SECONDARY OUTCOMES:
Any anti-tumor activity that may occur in patients receiving APX3330 using RECIST criteria | 18 months
  Using RECIST criteria

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - START Midwest, Grand Rapids, Michigan
  - START San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah F, Logsdon D, Messmann RA, Fehrenbacher JC, Fishel ML, Kelley MR. Exploiting the Ref-1-APE1 node in cancer signaling and other diseases: from bench to clinic. NPJ Precis Oncol. 2017;1:19. doi: 10.1038/s41698-017-0023-0. Epub 2017 Jun 8. PMID 28825044
- [Background] Jiang A, Gao H, Kelley MR, Qiao X. Inhibition of APE1/Ref-1 redox activity with APX3330 blocks retinal angiogenesis in vitro and in vivo. Vision Res. 2011 Jan;51(1):93-100. doi: 10.1016/j.visres.2010.10.008. Epub 2010 Oct 14. PMID 20937296
- [Result] Safi Shahda, Nehal J. Lakhani, Bert O'Neil, Drew W. Rasco, Jun Wan, Amber L Mosley, Hao Liu, Mark R. Kelley, Richard Adam Messmann. A phase I study of the APE1 protein inhibitor APX3330 in patients with advanced solid tumors. Journal of Clinical Oncology. Volume 37: Issue 15_suppl.
- [Derived] Kelley MR, Wan J, Liu S, Kpenu E, Wireman R, Mosley AL, Liu H, Lakhani NJ, Shahda S, O'Neil B, Opyrchal M, Messmann RA. A Phase I study targeting the APE1/ref-1 redox signaling protein with APX3330: First clinical agent targeting APE1/ref-1 in Cancer. Oncologist. 2025 Dec 19:oyaf423. doi: 10.1093/oncolo/oyaf423. Online ahead of print. PMID 41423797
- [Derived] Kelley MR, Wan J, Liu S, Kpenu E, Wireman R, Mosley AL, Liu H, Lakhani NJ, Shahda S, O'Neil B, Opyrchal M, Messmann RA. A Phase I study targeting the APE1/Ref-1 redox signaling protein with APX3330: First clinical agent targeting APE1/Ref-1 in Cancer. medRxiv [Preprint]. 2025 Apr 4:2025.04.03.25325173. doi: 10.1101/2025.04.03.25325173. PMID 40236444
- See also: Company website — http://apexianpharma.com